CLINICAL TRIAL: NCT02299310
Title: Effect of Valsartan vs Perindopril on HOMA-IR Index in Patients With Chronic Kidney Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ri-Bao Wei, Nephrology, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S2014-088
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease, Anti-hypertensive drugs
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Valsartan; lactitol; Perindopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valsartan (Experimental): Valsartan 80mg/tablet, 1 tablet once daily (crossover)
  Interventions: Drug: Valsartan
- Perindopril (Active Comparator): Perindopril 4mg/tablet, 1 tablet once daily (crossover)
  Interventions: Drug: Perindopril

INTERVENTIONS:
Drug: Valsartan — Valsartan 80mg/tablet, 1 tablet once daily (crossover)
  Other Names: NOVARTIS
  Arms: Valsartan
Drug: Perindopril — Perindopril 4mg/tablet, 1 tablet once daily (crossover)
  Other Names: ACERTIL
  Arms: Perindopril

SUMMARY:
The purpose of this study is to compare the effect of valsartan and perindopril on HOMA-IR Index in patients with chronic kidney disease.

DETAILED DESCRIPTION:
eligiable volunteers are administrated single-dose over the period I and II (crossover) of Valsartan (80mg) as of Perindopril (4mg).

Every time before and after each medication, HOMA-IR index and other parameters and safety of Valsartan (80mg) and Perindopril (4mg) is performed using a blood sample and conducting some tests (vital signs, physical exam, ECG, laboratory test, etc.) respectively.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic kidney disease
* Serum creatinine:1~3mg/dl

Exclusion Criteria:

* Diabetes
* Patients treated with corticosteroids or immunosuppressants
* BMI>30kg/m2
* SP>180mmHg, DP>110mmHg
* Patients with serious medical problems requiring specific medical treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Homeostasis model of assessment for insulin resistence index (HOMA-IR index) | 4 weeks
  HOMA-IR=FINS*FGLU/22.5

SECONDARY OUTCOMES:
Glomerular filtration rate(eGFR) and Creatinine clearance rate(CCR) | 4 weeks
  eGFR and CCR are calculated with MDRD formula
Body mass index(BMI) | 4 weeks
  BMI=weight/(height)^2
24-h urine protein, urinary albumin-creatinin ration, retinol binding protein | 4 weeks
Cholesterol, triglycerides, high density lipoprotein, low density lipoprotein | 4 weeks
Glycosylated hemoglobin | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: RiBao Wei, Master, Study Chair — Department of Nephrology, Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Satirapoj B, Leelasiri K, Supasyndh O, Choovichian P. Short-term administration of an angiotensin II receptor blocker in patients with long-term hemodialysis patients improves insulin resistance. J Med Assoc Thai. 2014 Jun;97(6):574-81. PMID 25137874
- [Background] Ushijima K, Takuma M, Ando H, Ishikawa-Kobayashi E, Nozawa M, Maekawa T, Shiga T, Fujimura A. Effects of telmisartan and valsartan on insulin sensitivity in obese diabetic mice. Eur J Pharmacol. 2013 Jan 5;698(1-3):505-10. doi: 10.1016/j.ejphar.2012.11.022. Epub 2012 Nov 27. PMID 23195328
- [Background] Iwashita M, Sakoda H, Kushiyama A, Fujishiro M, Ohno H, Nakatsu Y, Fukushima T, Kumamoto S, Tsuchiya Y, Kikuchi T, Kurihara H, Akazawa H, Komuro I, Kamata H, Nishimura F, Asano T. Valsartan, independently of AT1 receptor or PPARgamma, suppresses LPS-induced macrophage activation and improves insulin resistance in cocultured adipocytes. Am J Physiol Endocrinol Metab. 2012 Feb 1;302(3):E286-96. doi: 10.1152/ajpendo.00324.2011. Epub 2011 Nov 1. PMID 22045314